CLINICAL TRIAL: NCT01470599
Title: A Open-Label Extension Study Of CP-690,550 As Maintenance Therapy In Patients With Crohn's Disease
Brief Title: A Open-Label Study Of CP-690,550 As Long-Term Therapy (48 Weeks) In Subjects With Crohn's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A3921086; 2011-003622-27 (EudraCT Number)
Record Dates: First submitted 2011-10-27; First posted 2011-11-11 (Estimated); Results first posted 2017-10-16 (Actual); Last update posted 2017-10-16 (Actual); Status verified 2017-09

CONDITIONS: Crohn's Disease
MeSH Terms: conditions — Crohn Disease | interventions — tofacitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 5mg BID (Experimental)
  Interventions: Drug: CP-690,550
- 10mg BID (Experimental)
  Interventions: Drug: CP-690,550

INTERVENTIONS:
Drug: CP-690,550 — ORAL TABLET, TWICE DAILY
  Arms: 5mg BID
Drug: CP-690,550 — ORAL TABLETS, TWICE DAILY
  Arms: 10mg BID

SUMMARY:
The study hypothesis is to establish the safety and tolerability of long-term open-label (OL) CP-690,550 therapy in subjects with Crohn's disease.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who complete 26-week maintenance treatment of the A3921084 study or subjects who withdraw early due to A3921084 study treatment failure (see Appendix 5).
* Women of childbearing potential must test negative for pregnancy prior to study enrolment.
* Sexually active females of childbearing potential are required to use adequate contraceptive methods during the study period and until completion of the follow-up procedures. No specific contraceptive measures are required in male subjects during study participation.

Exclusion Criteria:

* Subjects who have been discontinued due to protocol violation(s) (as determined by the Sponsor) in the A3921084 study.
* Subjects who were discontinued from the A3921084 study due to an adverse event.
* Subjects likely to require any non-elective surgery or surgery requiring overnight stay (with the exception of minor same day outpatient procedures that will not interfere with study drug dosing).

Ages: 18 Years to 76 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2012-04 (Actual); Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (75):
- United States (32):
  - Alliance Clinical Research, Oceanside, California
  - Clinical Research Of The Rockies, Lafayette, Colorado
  - Gastroenterology Consultants of Clearwater, Clearwater, Florida
  - West Coast Endoscopy Center, Clearwater, Florida
  - Clinical Research of West Florida, Inc., Clearwater, Florida
  - Shands Endoscopy Center, Gainesville, Florida
  - Shands Hospital at the University of Florida, Gainesville, Florida
  - Investigational Drug Service, Gainesville, Florida
  - Shands Medical Plaza and Cancer Center, Gainesville, Florida
  - Gastroenterology Group of Naples, Naples, Florida
  - Gulfshore Endoscopy Center (Endoscopies Only), Naples, Florida
  - North Florida Gastroenterology Research, LLC, Orange Park, Florida
  - Internal Medicine Specialists, Orlando, Florida
  - Gastroenterology Associates of Central Georgia, LLC, Macon, Georgia
  - East Ann Arbor Health and Geriatrics Center, Ann Arbor, Michigan
  - University of Michigan Health Systems, Ann Arbor, Michigan
  - Center for Digestive Health, Troy, Michigan
  - Surgical Centers of Michigan, Troy, Michigan
  - NYU Langone Long Island Clinical Research Associates, Great Neck, New York
  - NYU Langone Nassau Gastroenterology Associates, Great Neck, New York
  - Cleveland Clinic, Cleveland, Ohio
  - Great Lakes Gastroenterology, Mentor, Ohio
  - The Endoscopy Center of Lake County, Mentor, Ohio
  - Great Lakes Gastroenterology, Willoughby, Ohio
  - Christus Trinity Mother Frances Endoscopy Center, Tyler, Texas
  - Digestive Health Specialists of Tyler, Tyler, Texas
  - Endoscopy Center of Tyler, Tyler, Texas
  - University of Utah HSC, Salt Lake City, Utah
  - Digestive and Liver Disease Specialists, Norfolk, Virginia
  - Wisconsin Center for Advanced Research - GI Associates, LLC, Milwaukee, Wisconsin
  - Allegiance Research Specialists, Wauwatosa, Wisconsin
  - GI Associates, Wauwatosa, Wisconsin
- Australia (3):
  - Nepean Public Hospital, Kingswood, New South Wales
  - Monash Medical Centre, Clayton, Victoria
  - Royal Melbourne Hospital, Parkville, Victoria
- AKH Wien Universitaetsklinik fuer Innere Medizin III, Vienna, Austria
- Bulgaria (2):
  - 4-MBAL, Parvo vatreshno otdelenie, Sofia
  - MBAL Sofiamed OOD, Otdelenie po gastroenterologia, Sofia
- Canada (5):
  - Office of Dr. David C Pearson, Victoria, British Columbia
  - Office of Drs. Ranjith Andrew Singh, Jamie D. Papp, Victoria, British Columbia
  - PerCuro Clinical Research Limited, Victoria, British Columbia
  - London Health Sciences Centre - University Hospital, London, Ontario
  - Montreal General Hospital-Mcgill University Health Centre, Montreal, Quebec
- Czechia (3):
  - Medial Pharma spol.s.r.o., Hradec Králové
  - RDG centrum s.r.o., Hradec Králové
  - Hepato-Gastroenterologie HK, s.r.o., Hradec Králové
- France (2):
  - Hopital Huriez - CHRU de Lille, Lille
  - Hôpital Haut-Lévêque, Pessac
- Germany (3):
  - Charite Universitaetsmedizin Berlin, Campus Benjamin Franklin, Berlin
  - Universitaetsklinikum Schleswig-Holstein, Kiel
  - Universitaetsklinikum Ulm, Ulm
- General Hospital of Athens "Evangelismos",1st Gastroenterology Department, Kolonaki Athens, Greece
- Hungary (5):
  - Peterfy Sandor Utcai Korhaz, Rendelointezet es Baleseti Kozpont, I. sz. Belgyogyaszat, Budapest
  - Pannonia Magánorvosi Centrum Kft, Budapest
  - Szent Janos Korhaz es Eszak-budai Egyesitett Korhazak, Budapest
  - Bugat Pal Korhaz Egeszsegugyi Szolgaltato Kozhasznu Nonprofit Kft.,, Gyöngyös
  - Clinfan Kft., Szekszárd
- Israel (3):
  - Department of medicine Shaare Zedek Medical Center, Jerusalem
  - Dept. of Gastroenterology & Hepatology, Meir Medical Center, Kfar Saba
  - Tel Aviv Sourasky Medical Center, Tel Aviv
- Japan (5):
  - Hokkaido P.W.F.A.C Sapporo-Kosei general Hospital, Sapporo, Hokkaido
  - The Hospital of Hyogo College of Medicine, Nishinomiya, Hyōgo
  - National Hospital Organization Sendai Medical Center, Sendai, Miyagi
  - Toho University Sakura Medical Center, Chiba
  - Osaka City University Hospital, Osaka
- Netherlands (2):
  - VU University Medical Center, Amsterdam
  - Academisch Medisch Centrum, Amsterdam
- Parklands Medical Centre, Durban, South Africa
- South Korea (2):
  - Samsung Medical Center, Seoul
  - Asan Medical Center, Soeul
- Spain (3):
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital Universitario de La Princesa, Madrid
  - Hospital Puerta de Hierro Majadahonda Servicio Digestivo - Planta 2, Madrid
- Ukraine (2):
  - Municipal Institution "Odesa Regional Clinical Hospital". Odesa Regional Centre of Gastroenterology., Odesa
  - Medical Clinical Research Center of Medical Center "Health Clinic" LLC, Vinnitsa

REFERENCES:
- [Derived] Panes J, D'Haens GR, Higgins PDR, Mele L, Moscariello M, Chan G, Wang W, Niezychowski W, Su C, Maller E. Long-term safety and tolerability of oral tofacitinib in patients with Crohn's disease: results from a phase 2, open-label, 48-week extension study. Aliment Pharmacol Ther. 2019 Feb;49(3):265-276. doi: 10.1111/apt.15072. PMID 30663107
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A3921086

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted in participants who completed the 26-week maintenance treatment of Study A3921084 or who withdrew early due to A3921084 study treatment failure according to prespecified criteria.
Pre-assignment Details: Participants were assigned to either the 5 milligram (mg) twice daily (BID) or 10 mg BID treatment group according to clinical remission status as assessed by Crohn's Disease Activity Index (CDAI) score at the end of the A3921084 study treatment visit or early termination visit due to A3921084 study treatment failure.
Groups:
- Tofacitinib 5 mg BID: Tofacitinib 5 mg tablet for oral administration at a dose of 5 mg BID for up to 48 weeks.
- Tofacitinib 10 mg BID: Tofacitinib 10 mg tablets (2 x 5 mg tablets) for oral administration at a dose of 10 mg BID for up to 48 weeks.
Period: Overall Study
Arm/Group | Tofacitinib 5 mg BID | Tofacitinib 10 mg BID
Started | 62 | 88
Completed | 43 | 45
Not Completed | 19 | 43
Not completed — Did not meet entrance criteria | 1 | 0
Not completed — Lost to Follow-up | 2 | 1
Not completed — Withdrawal by Subject | 3 | 4
Not completed — Other | 1 | 0
Not completed — Protocol Violation | 3 | 1
Not completed — Adverse event related to study drug | 2 | 5
Not completed — Insufficient clinical response | 6 | 27
Not completed — Adverse event not related to study drug | 1 | 5

BASELINE CHARACTERISTICS:
Population: The safety analysis set (SAS) consisted of all participants enrolled in this open label (OL) extension study who received at least 1 dose of study medication.
Groups:
- Total: Total of all reporting groups
Arm/Group | Tofacitinib 5 mg BID | Tofacitinib 10 mg BID | Total
Number analyzed (Participants) | 62 | 88 | 150
Age, Continuous [Mean (Standard Deviation); unit: Years] | 41.0 (12.6) | 38.2 (11.6) | 39.4 (12.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 41 | 71
  Male | 32 | 47 | 79

OUTCOME MEASURES:

1. Primary Outcome: Adjudicated Potential Cardiovascular Events
Description: Pre-specified cardiovascular events were adjudicated by committees of external experts who were blinded to treatment assignment. Potential events of interest (pEoI) were identified by the investigator, sponsor, review of alerts from central electrocardiogram assessments, and by search of adverse events (AE)/serious adverse event (SAE) listings for events coded to death (coronary and non-coronary), myocardial infarction (non-fatal), all coronary revascularization, unstable angina, stroke (fatal and non-fatal), transient ischemic attack, congestive heart failure, peripheral arterial vascular disease, dyspnoea, and chest pain. The independent reviewers (IRs) determined if the pEoI met the criteria for EoI classification according to the definitions summarized from the Clinical Data Interchange Standards Consortium 'Standardized Definitions for End Point Events in Cardiovascular Trials' published October 2010.
Time Frame: From baseline to Week 52
Population: Participants in the SAS who had pEoI and were adjudicated by IRs
Measure: Number; unit: Number of events meeting criteria
Arm/Group | Tofacitinib 5 mg BID | Tofacitinib 10 mg BID
Number analyzed (Participants) | 0 | 2
Number of events meeting criteria |  | 0

2. Primary Outcome: Adjudicated Malignancy Events
Description: Pre-specified malignancy events were adjudicated by committees of external experts who were blinded to treatment assignment. pEoI were identified by the investigator, sponsor, potential primary event notifications (i.e. malignancies excluding non-melanoma skin cancers) for a specific protocol, events submitted for histopathology review for potential malignancies which met the criteria for potential malignancies, and by search of AE/SAE listings for events coded to Malignant tumors Standard Medical Dictionary for Regulatory Activities (MedDRA) Queries (SMQ) (20000194). IRs determined if the pEoI met the criteria for EoI classification according to the International Classification of Diseases for Oncology, a ten-digit multi-axial classification of the site (4 characters), morphology (4 digits), behavior (1 digit), and grading (1 digit) of neoplasms.
Time Frame: From baseline to Week 52
Population: Participants in the SAS who had pEoI and were adjudicated by IRs
Measure: Number; unit: Number of events meeting criteria
Arm/Group | Tofacitinib 5 mg BID | Tofacitinib 10 mg BID
Number analyzed (Participants) | 1 | 1
Number of events meeting criteria | 0 | 1

3. Secondary Outcome: Percentage of Participants in Clinical Remission and Sustained Clinical Remission at Week 48
Description: CDAI is a composite index consisting of weighted scoring of 8 disease variables: number of liquid or very soft stools, intensity of abdominal pain, general well-being, occurrence of extraintestinal symptoms, need for antidiarrheal drugs, presence of abdominal masses, hematocrit, and body weight. CDAI scores range from 0 to approximately 600 points, higher score indicates higher disease activity. Clinical remission was defined as a CDAI score of less than (<) 150. Sustained clinical remission was defined as being in clinical remission (CDAI score <150) at both Week 24 and Week 48. 95 percent (%) Clopper-Pearson exact confidence interval reported for the proportions. n = number of participants with non-missing data.
Time Frame: Week 48
Population: Full analysis set (FAS) - consisted of all participants enrolled in this OL extension study.
Measure: Number (95% Confidence Interval); unit: Percent
Arm/Group | Tofacitinib 5 mg BID | Tofacitinib 10 mg BID
Number analyzed (Participants) | 62 | 88
Percent
  Clinical remission (n=33, 36) | 87.88 [71.80 to 96.60] | 55.56 [38.10 to 72.06]
  Sustained clinical remission (n=32, 35) | 75.00 [56.60 to 88.54] | 34.29 [19.13 to 52.21]

4. Secondary Outcome: Percentage of Participants in Clinical Remission and Sustained Clinical Remission Among Participants in Clinical Remission at Baseline of This Study
Description: CDAI is a composite index consisting of weighted scoring of 8 disease variables: number of liquid or very soft stools, intensity of abdominal pain, general well-being, occurrence of extraintestinal symptoms, need for antidiarrheal drugs, presence of abdominal masses, hematocrit, and body weight. CDAI scores range from 0 to approximately 600 points, higher score indicates higher disease activity. Clinical remission was defined as a CDAI score of <150. Sustained clinical remission was defined as being in clinical remission (CDAI score <150) at both Week 24 and Week 48. 95% Clopper-Pearson exact confidence interval reported for the proportions. n = number of participants with non-missing data.
Time Frame: Baseline and Weeks 8, 16, 24, 36, 48 and 52/follow-up
Population: Participants in the FAS who met clinical remission criteria at baseline of this study
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Tofacitinib 5 mg BID | Tofacitinib 10 mg BID
Number analyzed (Participants) | 61 | 4
Percentage of participants
  Clinical remission: Baseline (n=61, 4) | 100.00 [94.13 to 100.00] | 100.00 [39.76 to 100.00]
  Clinical remission: Week 8 (n=53, 4) | 75.47 [61.72 to 86.24] | 50.00 [6.76 to 93.24]
  Clinical remission: Week 16 (n=52, 4) | 84.62 [71.92 to 93.12] | 75.00 [19.41 to 99.37]
  Clinical remission: Week 24 (n=48, 4) | 85.42 [72.24 to 93.93] | 25.00 [0.63 to 80.59]
  Clinical remission: Week 36 (n=40, 3) | 92.50 [79.61 to 98.43] | 33.33 [0.84 to 90.57]
  Clinical remission: Week 48 (n=32, 3) | 87.50 [71.01 to 96.49] | 100.00 [29.24 to 100.00]
  Clinical remission: Week 52/follow-up (n=37, 3) | 64.86 [47.46 to 79.79] | 33.33 [0.84 to 90.57]
  Sustained clinical remission (n=31, 3) | 77.42 [58.90 to 90.41] | 33.33 [0.84 to 90.57]

5. Secondary Outcome: Percentage of Participants in Clinical Remission and Sustained Clinical Remission Among Participants in Clinical Response (CDAI-100 Response) or Clinical Remission at Baseline of This Study
Description: CDAI is a composite index consisting of weighted scoring of 8 disease variables: number of liquid or very soft stools, intensity of abdominal pain, general well-being, occurrence of extraintestinal symptoms, need for antidiarrheal drugs, presence of abdominal masses, hematocrit, and body weight. CDAI scores range from 0 to approximately 600 points, higher score indicates higher disease activity. Clinical remission was defined as a CDAI score of <150. Sustained clinical remission was defined as being in clinical remission (CDAI score <150) at both Week 24 and Week 48. Clinical response was defined as a CDAI score reduction of at least 100 points from the A3921083 study baseline value. 95% Clopper-Pearson exact confidence interval reported for the proportions. n = number of participants with non-missing data.
Time Frame: Baseline and Weeks 8, 16, 24, 36, 48 and 52/follow-up
Population: Participants in the FAS who met clinical response or clinical remission criteria at baseline of this study
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Tofacitinib 5 mg BID | Tofacitinib 10 mg BID
Number analyzed (Participants) | 62 | 23
Percentage of participants
  Clinical remission: Baseline (n=62, 23) | 98.39 [91.34 to 99.96] | 17.39 [4.95 to 38.78]
  Clinical remission: Week 8 (n=54, 20) | 75.93 [62.36 to 86.51] | 35.00 [15.39 to 59.22]
  Clinical remission: Week 16 (n=53, 19) | 84.91 [72.41 to 93.25] | 36.84 [16.29 to 61.64]
  Clinical remission: Week 24 (n=49, 16) | 83.67 [70.34 to 92.68] | 43.75 [19.75 to 70.12]
  Clinical remission: Week 36 (n=41, 13) | 90.24 [76.87 to 97.28] | 38.46 [13.86 to 68.42]
  Clinical remission: Week 48 (n=33, 10) | 87.88 [71.80 to 96.60] | 50.00 [18.71 to 81.29]
  Clinical remission: Week 52/follow-up (n=38, 12) | 65.79 [48.65 to 80.37] | 41.67 [15.17 to 72.33]
  Sustained clinical remission (n=32, 10) | 75.00 [56.60 to 88.54] | 30.00 [6.67 to 62.25]

6. Secondary Outcome: Time to Relapse Among Participants in Clinical Remission at Baseline
Description: Relapse was defined as an increase in CDAI of more than (>) 100 points from the baseline and an absolute CDAI score of >220 points. CDAI is a composite index consisting of weighted scoring of 8 disease variables: number of liquid or very soft stools, intensity of abdominal pain, general well-being, occurrence of extraintestinal symptoms, need for antidiarrheal drugs, presence of abdominal masses, hematocrit, and body weight. CDAI scores range from 0 to approximately 600 points, higher score indicates higher disease activity. Data presented are rates estimated from Kaplan-Meier curves.
  n = number of participants remaining at risk.
Time Frame: From baseline to Week 52
Population: Participants in the FAS who met clinical remission criteria at baseline of this study
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Tofacitinib 5 mg BID | Tofacitinib 10 mg BID
Number analyzed (Participants) | 61 | 4
Percentage of participants
  Week 8 (n=55, 4) | 6.78 [3.38 to 11.78] | NA [NA to NA] — No participants had a relapse event by Week 8.
  Week 16 (n=51, 3) | 11.86 [7.15 to 17.87] | 25.00 [4.56 to 53.66]
  Week 24 (n=46, 3) | 15.46 [9.98 to 22.05] | 25.00 [4.56 to 53.66]
  Week 36 (n=38, 3) | 21.42 [14.82 to 28.83] | 25.00 [4.56 to 53.66]
  Week 48 (n=7, 0) | 24.69 [17.21 to 32.89] | NA [NA to NA] — No participants remained at risk of a relapse event by Week 48.

7. Secondary Outcome: Observed CDAI Score by Week
Description: CDAI is a composite index consisting of weighted scoring of 8 disease variables: number of liquid or very soft stools, intensity of abdominal pain, general well-being, occurrence of extraintestinal symptoms, need for antidiarrheal drugs, presence of abdominal masses, hematocrit, and body weight. CDAI scores range from 0 to approximately 600 points, higher score indicates higher disease activity. n = number of participants remaining at risk.
Time Frame: Baseline and Weeks 8, 16, 24, 36, 48 and 52/follow-up
Population: FAS
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Tofacitinib 5 mg BID | Tofacitinib 10 mg BID
Number analyzed (Participants) | 62 | 88
Score on a scale
  Baseline (n=62, 88) | 77.13 (43.22) | 291.19 (95.78)
  Week 8 (n=54, 75) | 105.39 (75.82) | 176.96 (82.39)
  Week 16 (n=53, 66) | 86.58 (65.23) | 178.94 (72.25)
  Week 24 (n=49, 59) | 85.12 (56.67) | 163.66 (79.73)
  Week 36 (n=41, 48) | 73.34 (59.52) | 158.67 (89.15)
  Week 48 (n=33, 36) | 73.91 (70.23) | 154.11 (71.47)
  Week 52/Follow-up (n=38, 43) | 129.32 (114.82) | 180.65 (98.80)

8. Secondary Outcome: Change From Baseline Observed CDAI Score by Week
Description: CDAI is a composite index consisting of weighted scoring of 8 disease variables: number of liquid or very soft stools, intensity of abdominal pain, general well-being, occurrence of extraintestinal symptoms, need for antidiarrheal drugs, presence of abdominal masses, hematocrit, and body weight. CDAI scores range from 0 to approximately 600 points, higher score indicates higher disease activity. n = number of participants with non-missing data.
Time Frame: Weeks 8, 16, 24, 36, 48 and 52/follow-up
Population: FAS
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Tofacitinib 5 mg BID | Tofacitinib 10 mg BID
Number analyzed (Participants) | 62 | 88
Score on a scale
  Week 8 (n=54, 75) | 26.96 (62.68) | -114.31 (112.44)
  Week 16 (n=53, 66) | 11.72 (52.25) | -112.02 (111.09)
  Week 24 (n=49, 59) | 6.33 (44.48) | -122.69 (117.65)
  Week 36 (n=41, 48) | -10.78 (40.35) | -139.81 (126.18)
  Week 48 (n=33, 36) | -4.79 (60.09) | -121.94 (129.21)
  Week 52/Follow-up (n=38, 43) | 47.66 (109.73) | -107.42 (119.05)

9. Secondary Outcome: Percentage of Participants Achieving a Steroid-Free Clinical Remission at Week 48 - Among Subjects on Steroids at A3921086 Baseline
Description: Steroid-free clinical remission at Week 48 was a CDAI <150 points in participants who were steroid-free at Week 48. CDAI is a composite index consisting of weighted scoring of 8 disease variables: number of liquid or very soft stools, intensity of abdominal pain, general well-being, occurrence of extraintestinal symptoms, need for antidiarrheal drugs, presence of abdominal masses, hematocrit, and body weight. CDAI scores range from 0 to approximately 600 points, higher score indicates higher disease activity.
Time Frame: Week 48
Population: Participants in FAS who were on steroids at baseline of this study
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Tofacitinib 5 mg BID | Tofacitinib 10 mg BID
Number analyzed (Participants) | 2 | 11
Percentage of participants | 50.00 [1.26 to 98.74] | 9.09 [0.23 to 41.28]

10. Secondary Outcome: Corticosteroid Use Over Time
Description: Use of corticosteroids (yes or no) was recorded at baseline and throughout the study. Percentage of participants taking corticosteriod at each visit was reported.
Time Frame: Weeks 8, 16, 24, 36 and 48
Population: SAS
Measure: Number; unit: Percentage of participants
Arm/Group | Tofacitinib 5 mg BID | Tofacitinib 10 mg BID
Number analyzed (Participants) | 62 | 88
Percentage of participants
  Baseline | 1.61 | 20.45
  Week 8 | 4.84 | 21.59
  Week 16 | 4.84 | 13.64
  Week 24 | 4.84 | 12.50
  Week 36 | 3.23 | 10.23
  Week 48 | 1.61 | 7.95

11. Secondary Outcome: Percentage of Participants Switching From 5 mg BID to 10 mg BID or 10 mg BID to 5 mg BID After Initial Assignment by Visit
Description: There was a single study treatment dose adjustment allowed, at the discretion of the Investigator, from 5 mg BID to 10 mg BID or from 10 mg BID to 5 mg BID, after the initial 8 weeks of fixed open label treatment and for the remaining treatment period of 40 weeks. Percentage of participants whose study treatment were switched from 5 mg BID to 10 mg BID or 10 mg BID to 5 mg BID after initial assignment was reported.
Time Frame: From baseline to Week 48
Population: FAS
Measure: Number; unit: Percentage of participants
Arm/Group | Tofacitinib 5 mg BID | Tofacitinib 10 mg BID
Number analyzed (Participants) | 62 | 88
Percentage of participants
  Baseline | 0 [0.00 to 5.78] | 0 [0.00 to 4.11]
  Week 8 | 25.81 [15.53 to 38.50] | 0 [0.00 to 4.11]
  Week 16 | 6.45 [1.79 to 15.70] | 0 [0.00 to 4.11]
  Week 24 | 3.23 [0.39 to 11.71] | 2.27 [0.28 to 7.97]
  Week 36 | 0 [0.00 to 5.78] | 1.14 [0.03 to 6.17]
  Week 48 | 0 [0.00 to 5.78] | 0 [0.00 to 4.11]

12. Secondary Outcome: Observed Change From Baseline in Fecal Calprotectin by Week
Description: Fecal calprotectin is an inflammatory marker for the gastrointestinal tract and considered as a measurement of neutrophil migration to the gastrointestinal tract. Higher values indicate more serious inflammation. n = number of participants with non-missing data.
Time Frame: Baseline and Weeks 8, 16, 24, 36, 48 and 52/follow-up
Population: FAS
Measure: Mean (Standard Deviation); unit: mg per kilogram (mg/kg)
Arm/Group | Tofacitinib 5 mg BID | Tofacitinib 10 mg BID
Number analyzed (Participants) | 62 | 88
mg per kilogram (mg/kg)
  Week 8 (n=53, 71) | -105.51 (436.41) | -102.82 (310.10)
  Week 16 (n=54, 64) | -144.65 (423.20) | -35.28 (718.82)
  Week 24 (n=49, 55) | -120.49 (511.49) | -130.68 (337.23)
  Week 36 (n=41, 42) | -169.92 (354.30) | -133.82 (364.51)
  Week 48 (n=37, 38) | -189.61 (462.61) | -123.87 (376.70)
  Week 52/Follow-up (n=48, 57) | -51.33 (453.73) | -109.23 (389.54)

13. Secondary Outcome: Observed Change From Baseline in High Sensitivity C-reactive Protein (CRP) by Week
Description: The test for CRP is a laboratory measurement for evaluation of an acute phase reactant of inflammation through the use of an ultrasensitive assay. A decrease in the level of CRP indicates reduction in inflammation and therefore improvement. n = number of participants with non-missing data.
Time Frame: Baseline and Weeks 8, 16, 24, 36, 48 and 52/follow-up
Population: FAS
Measure: Mean (Standard Deviation); unit: mg per liter (mg/L)
Arm/Group | Tofacitinib 5 mg BID | Tofacitinib 10 mg BID
Number analyzed (Participants) | 62 | 88
mg per liter (mg/L)
  Week 8 (n=61, 82) | -0.44 (14.78) | -4.81 (26.76)
  Week 16 (n=58, 72) | -2.46 (14.54) | -7.96 (25.11)
  Week 24 (n=54, 61) | -2.76 (17.59) | -9.26 (30.20)
  Week 36 (n=46, 51) | -4.42 (22.29) | -12.09 (30.61)
  Week 48 (n=43, 44) | -4.55 (17.81) | -11.45 (31.30)
  Week 52/Follow-up (n=54, 71) | 3.86 (21.57) | -4.72 (31.34)

14. Secondary Outcome: Inflammatory Bowel Disease Questionnaire (IBDQ) Total Score and Domain Scores (Bowel Function, Emotional Status, Systemic Symptoms, and Social Function) at Baseline and Week 48/ET Visit
Description: The IBDQ is a psychometrically validated patient reported outcome (PRO) instrument for measuring disease-specific quality of life (QoL) in participants with inflammatory bowel disease (IBD). IBDQ consists of 32 items, each item score ranged from 1 (worst possible response) to 7 (best possible response). The 32 items are grouped into 4 domains: bowel function, emotional status, systemic symptoms and social function. The 4 domains are scored as follows: bowel symptoms 10 to 70; systemic symptoms 5 to 35; emotional function 12 to 84; social function 5 to 35. For each domain, a higher score indicates better QoL. Total score is the sum of each item score, and ranged from 32 to 224 with a higher score indicating a better QoL. Positive change in total score indicated improvement in QoL. n = number of participants with non-missing data.
Time Frame: Baseline and Week 48/early termination (ET)
Population: FAS
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Tofacitinib 5 mg BID | Tofacitinib 10 mg BID
Number analyzed (Participants) | 62 | 88
Score on a scale
  IBDQ Total Score, Baseline (n=62, 87) | 187.23 (20.38) | 127.32 (34.17)
  IBDQ Total Score, Week 48/ET (n=57, 83) | 179.26 (29.89) | 144.42 (42.16)
  Bowel Function Score, Baseline (n=62, 87) | 58.56 (6.86) | 40.71 (9.90)
  Bowel Function Score, Week 48/ET (n=57, 83) | 55.70 (9.82) | 46.70 (12.38)
  Emotional Status Score, Baseline (n=62, 87) | 69.68 (8.58) | 48.61 (14.42)
  Emotional Status Score, Week 48/ET (n=57, 83) | 66.98 (12.27) | 53.19 (17.32)
  Systemic Symptoms Score, Baseline (n=62, 87) | 26.95 (5.36) | 17.20 (5.55)
  Systemic Symptoms Score, Week 48/ET (n=57, 83) | 25.82 (6.28) | 20.35 (7.07)
  Social Function Score, Baseline (n=62, 87) | 32.03 (3.59) | 20.80 (8.96)
  Social Function Score, Week 48/ET (n=57, 83) | 30.75 (5.17) | 24.18 (8.98)

15. Secondary Outcome: Change From Baseline IBDQ Total Score and Domain Scores (Bowel Function, Emotional Status, Systemic Symptoms, and Social Function) at Week 48/ET Visit
Description: The IBDQ is a psychometrically validated PRO instrument for measuring disease-specific QoL in participants with IBD. IBDQ consists of 32 items, each item score ranged from 1 (worst possible response) to 7 (best possible response). The 32 items are grouped into 4 domains: bowel function, emotional status, systemic symptoms and social function. The 4 domains are scored as follows: bowel symptoms 10 to 70; systemic symptoms 5 to 35; emotional function 12 to 84; social function 5 to 35. For each domain, a higher score indicates better QoL. Total score is the sum of each item score, and ranged from 32 to 224 with a higher score indicating a better QoL. Positive change in total score indicated improvement in QoL.
Time Frame: Baseline and Week 48/ET
Population: Participants in the FAS who had non-missing data at Week 48/ET visit
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Tofacitinib 5 mg BID | Tofacitinib 10 mg BID
Number analyzed (Participants) | 57 | 83
Score on a scale
  IBDQ Total Score, Week 48/ET | -7.98 (24.93) | 18.84 (40.45)
  Bowel Function Score, Week 48/ET | -2.72 (8.30) | 6.37 (12.41)
  Emotional Status Score, Week 48/ET | -3.07 (10.48) | 5.36 (15.00)
  Systemic Symptoms Score, Week 48/ET | -1.00 (4.83) | 3.45 (7.43)
  Social Function Score, Week 48/ET | -1.19 (4.24) | 3.66 (8.89)

16. Secondary Outcome: Percentage of Participants With an IBDQ Total Score of Greater Than or Equal to (≥) 170 at Week 48/ET Visit
Description: The IBDQ is a psychometrically validated PRO instrument for measuring disease-specific QoL in participants with IBD. IBDQ consists of 32 items, each item score ranged from 1 (worst possible response) to 7 (best possible response). Total score is the sum of each item score, and ranged from 32 to 224 with a higher score indicating a better QoL. A score ≥170 corresponds to clinical remission. 95% Clopper-Pearson exact confidence interval reported for the proportions.
Time Frame: Week 48/ET
Population: Participants in the FAS who had non-missing data at Week 48/ET visit
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Tofacitinib 5 mg BID | Tofacitinib 10 mg BID
Number analyzed (Participants) | 57 | 83
Percentage of participants | 70.18 [56.60 to 81.57] | 31.33 [21.59 to 42.44]

17. Secondary Outcome: Percentage of Participants With a Response to the Patient-Reported Treatment Impact (PRTI) Assessment at Week 48/ET Visit by Category
Description: The IBD PRTI modified questionnaire comprises 3 individual questions administered to the participant: participant satisfaction with study treatment; participant preference for study drug over prior treatment (this question on participant preference for study drug is prefaced by a simple question of previous treatment/s for IBD received in order to place the preference question into context) and participant willingness to reuse the study treatment again. Each of these questions (except the question on previous treatment, which is informational only) is scored on a 5 point Likert scale. PSA = Patient Satisfaction Assessment; PPTA = Patient Previous Treatment Assessment; PPA = Patient Preference Assessment; PWA = Patient Willingness Assessment.
Time Frame: Week 48/ET visit
Population: Participants in the FAS who had a response to PRTI assessment at Week 48/ET visit
Measure: Number; unit: Percentage of participants
Arm/Group | Tofacitinib 5 mg BID | Tofacitinib 10 mg BID
Number analyzed (Participants) | 42 | 46
Percentage of participants
  PSA: Extremely dissatisfied | 0 | 0
  PSA: Dissatisfied | 0 | 8.7
  PSA: Neither satisfied nor dissatisfied | 0 | 17.4
  PSA: Satisfied | 33.3 | 41.3
  PSA: Extremely satisfied | 66.7 | 32.6
  PPTA: Injectable prescription medicines | 40.5 | 32.6
  PPTA: Prescription medicines taken by mouth | 45.2 | 43.5
  PPTA: Surgery | 2.4 | 0
  PPTA: Prescription medicines & surgery | 7.1 | 13.0
  PPTA: No treatment | 4.8 | 10.9
  PPA: Definitely prefer the drug I am receiving now | 88.1 | 56.5
  PPA: Slight preference for drug I'm receiving now | 4.8 | 21.7
  PPA: I have no preference either way | 7.1 | 17.4
  PPA: Slight preference for previous treatment | 0 | 4.3
  PPA: No, I definitely prefer my previous treatment | 0 | 0
  PWA: Would definitely want to use same drug again | 83.3 | 60.9
  PWA: Might want to use the same drug again | 14.3 | 23.9
  PWA: I am not sure | 2.4 | 10.9
  PWA: Might not want to use same drug again | 0 | 0
  PWA: Definitely not want to use same drug again | 0 | 4.3

18. Secondary Outcome: Short Form 36 Health Survey (SF-36) Component and Domain Scores at Baseline and Week 48/ET Visit
Description: The component and domain scores were scored using the United States (US) 1998 general population norms. The resulting norm-based T scores for both the SF36 version 2 and SF36 health domain scales and component summary measures have means of 50 and standard deviations of 10. Higher scores indicate better health-related QoL. n = number of participants with non-missing data.
Time Frame: Baseline and Week 48/ET visit
Population: FAS
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Tofacitinib 5 mg BID | Tofacitinib 10 mg BID
Number analyzed (Participants) | 62 | 88
Score on a scale
  Physical component score, Baseline (n=62, 86) | 50.15 (6.73) | 37.80 (9.53)
  Physical component score, Week 48/ET (n=57, 83) | 48.43 (8.22) | 41.87 (10.06)
  Mental Component Score, Baseline (n=62, 86) | 50.25 (9.11) | 37.17 (11.94)
  Mental Component Score, Week 48/ET (n=57, 83) | 48.79 (10.64) | 39.60 (12.87)
  Physical Functioning Domain, Baseline (n=62, 86) | 53.35 (5.50) | 43.50 (10.37)
  Physical Functioning Domain, Week 48/ET (n=57, 83) | 51.40 (8.59) | 46.81 (10.22)
  Role Physical Domain, Baseline (n=62, 86) | 50.97 (8.22) | 35.93 (11.30)
  Role Physical Domain, Week 48/ET (n=57, 83) | 49.38 (8.78) | 40.04 (12.99)
  Bodily Pain Domain, Baseline (n=62, 87) | 51.32 (8.55) | 35.31 (9.14)
  Bodily Pain Domain, Week 48/ET (n=57, 83) | 49.57 (10.30) | 41.04 (12.69)
  General Health Domain, Baseline (n=62, 87) | 41.60 (9.51) | 31.74 (8.41)
  General Health Domain, Week 48/ET (n=57, 83) | 40.39 (10.08) | 33.45 (10.16)
  Vitality Domain, Baseline (n=62, 87) | 52.78 (10.68) | 36.92 (9.88)
  Vitality Domain, Week 48/ET (n=57, 83) | 51.06 (11.38) | 41.03 (12.38)
  Social Functioning Domain, Baseline (n=62, 87) | 51.81 (7.21) | 36.38 (12.29)
  Social Functioning Domain, Week 48/ET (n=57, 83) | 49.42 (9.64) | 39.82 (13.39)
  Role Emotional Domain, Baseline (n=62, 86) | 50.12 (8.85) | 38.55 (12.73)
  Role Emotional Domain, Week 48/ET (n=57, 83) | 47.97 (10.78) | 41.13 (13.15)
  Mental Health Domain, Baseline (n=62, 87) | 49.89 (9.84) | 37.61 (11.98)
  Mental Health Domain, Week 48/ET (n=57, 83) | 49.24 (10.27) | 40.13 (12.52)

19. Secondary Outcome: Change From Baseline SF-36 Component and Domain Scores at Week 48/ET Visit
Description: The component and domain scores were scored using the US 1998 general population norms. The resulting norm-based T scores for both the SF36 version 2 and SF36 health domain scales and component summary measures have means of 50 and standard deviations of 10. Higher scores indicate better health-related QoL. n = number of participants with non-missing data.
Time Frame: Baseline and Week 48/ET visit
Population: FAS
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Tofacitinib 5 mg BID | Tofacitinib 10 mg BID
Number analyzed (Participants) | 62 | 88
Score on a scale
  Physical component score, Week 48/ET (n=57, 83) | -1.47 (7.17) | 4.47 (11.06)
  Mental Component Score, Week 48/ET (n=57, 83) | -1.88 (9.05) | 3.07 (11.53)
  Physical Functioning Domain, Week 48/ET (n=57, 83) | -1.80 (7.50) | 3.49 (10.74)
  Role Physical Domain, Week 48/ET (n=57, 83) | -1.38 (7.87) | 4.60 (12.62)
  Bodily Pain Domain, Week 48/ET (n=57, 83) | -1.60 (7.90) | 6.15 (12.92)
  General Health Domain, Week 48/ET (n=57, 83) | -1.42 (10.00) | 2.25 (7.99)
  Vitality Domain, Week 48/ET (n=57, 83) | -1.63 (10.39) | 4.47 (12.16)
  Social Functioning Domain, Week 48/ET (n=57, 83) | -2.92 (9.09) | 3.69 (13.46)
  Role Emotional Domain, Week 48/ET (n=57, 82) | -2.26 (10.29) | 3.28 (11.38)
  Mental Health Domain, Week 48/ET (n=57, 83) | -1.02 (8.63) | 2.87 (11.72)

20. Secondary Outcome: EuroQoL 5 Dimensions Questionnaire (EQ-5D) Utility Scores at Baseline and Week 48/ET Visit
Description: EQ5D is a participant rated questionnaire to assess health-related QoL in terms of a single utility score. Health State Profile component assesses level of current health for 5 domains: mobility, selfcare, usual activities, pain and discomfort, and anxiety and depression; 1 indicates better health state (no problems); 3 indicates worst health state ("confined to bed"). Scoring formula developed by EuroQol Group assigns a utility value for each domain in the profile. Score is transformed and results in a total score range from 0.594 to 1.000; a higher score indicates a better health state. n = number of participants with non-missing data.
Time Frame: Baseline and Week 48/ET visit
Population: FAS
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Tofacitinib 5 mg BID | Tofacitinib 10 mg BID
Number analyzed (Participants) | 62 | 88
Score on a scale
  Utility Score, Baseline (n=62, 85) | 0.85 (0.21) | 0.57 (0.28)
  Utility Score, Week 48/ET (n=57, 83) | 0.84 (0.16) | 0.66 (0.31)

21. Secondary Outcome: Change From Baseline EQ-5D Utility Scores at Week 48/ET Visit
Description: EQ5D is a participant rated questionnaire to assess health-related QoL in terms of a single utility score. Health State Profile component assesses level of current health for 5 domains: mobility, selfcare, usual activities, pain and discomfort, and anxiety and depression; 1 indicates better health state (no problems); 3 indicates worst health state ("confined to bed"). Scoring formula developed by EuroQol Group assigns a utility value for each domain in the profile. Score is transformed and results in a total score range from 0.594 to 1.000; a higher score indicates a better health state.
Time Frame: Baseline and Week 48/ET visit
Population: Participants in the FAS who had non-missing data at Week 48/ET visit
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Tofacitinib 5 mg BID | Tofacitinib 10 mg BID
Number analyzed (Participants) | 57 | 83
Score on a scale | -0.02 (0.21) | 0.10 (0.36)

22. Secondary Outcome: EQ-5D Visual Analogue Scale (VAS) Scores at Baseline and Week 8/ET Visit
Description: EQ5D is a participant rated questionnaire to assess health-related QoL in terms of a single index value. The VAS component rates current health state on a scale from 0 millimeters (mm) (worst imaginable health state) to 100 mm (best imaginable health state); higher scores indicate a better health state. n = number of participants with non-missing data.
Time Frame: Baseline and Week 48/ET visit
Population: FAS
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Tofacitinib 5 mg BID | Tofacitinib 10 mg BID
Number analyzed (Participants) | 62 | 88
mm
  VAS Score, Baseline (n=62, 86) | 77.98 (16.18) | 48.60 (19.21)
  VAS Score, Week 48/ET (n=57, 83) | 73.40 (18.54) | 57.60 (24.60)

23. Secondary Outcome: Change From Baseline EQ-5D VAS Scores at Week 8/ET Visit
Description: EQ5D is a participant rated questionnaire to assess health-related QoL in terms of a single index value. The VAS component rates current health state on a scale from 0 mm (worst imaginable health state) to 100 mm (best imaginable health state); higher scores indicate a better health state.
Time Frame: Baseline and Week 48/ET visit
Population: Participants in the FAS who had non-missing data at Week 48/ET visit
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Tofacitinib 5 mg BID | Tofacitinib 10 mg BID
Number analyzed (Participants) | 57 | 83
mm | -3.79 (20.56) | 10.16 (26.57)

24. Secondary Outcome: Percentage of Participants Hospitalized Due to Crohn's Disease
Description: The number of participants hospitalized due to Crohn's disease were recorded at every study visit.
Time Frame: From baseline to Week 52/follow-up
Population: SAS
Measure: Number; unit: Percentage of participants
Arm/Group | Tofacitinib 5 mg BID | Tofacitinib 10 mg BID
Number analyzed (Participants) | 62 | 88
Percentage of participants | 11.3 | 15.9

25. Primary Outcome: Adjudicated Hepatic Injury Events
Description: Pre-specified liver injury events were adjudicated by blinded committees of external experts. pEoI were identified by investigator, sponsor & search of clinical, safety & laboratory databases (potential Hy's law event, ALT/AST ≥5 x ULN, events meeting hepatic discontinuation criteria, SAEs coded to MedDRA hepatobiliary system organ class (SOC), AEs/SAEs coded to MedDRA liver infections or infectious biliary disorders SMQ, AEs coded to MedDRA drug-induced liver injury (DILI) preferred term or any death with ALT or AST ≥3xULN, bilirubin ≥2xULN or jaundice). IRs determined if the pEoI met the criteria for EoI classification by assessing DILI (definite, highly likely, probable, possible, unlikely, unrelated or undetermined), pattern (hepatocellular, mixed, cholestatic or undetermined), likely, competing or alternative cause(s), severity (mild, moderate, severe, fatal/transplantation or undetermined), Hy's law case, recovery & liver failure (all yes, no or undetermined).
Time Frame: From baseline to Week 52
Population: Participants in the SAS who had pEoI and were adjudicated by IRs
Measure: Number; unit: Number of events meeting criteria
Arm/Group | Tofacitinib 5 mg BID | Tofacitinib 10 mg BID
Number analyzed (Participants) | 0 | 1
Number of events meeting criteria |  | 0

26. Primary Outcome: Adjudicated Opportunistic Infection Events
Description: Pre-specified opportunistic infection events were adjudicated by blinded committees of external experts. pEoI were identified by investigator, sponsor & search of SAE listings for serious infections coded to MedDRA infections & infestations SOC &/or events meeting pre-specified criteria for IR pre-screening to determine if adjudication is required. IRs determined if the pEoI met the criteria for EoI classification according to definitions for opportunistic infections (invasive fungal infections per the European Organization for Research & Treatment of Cancer/Invasive Fungal Infections Cooperative Group & the National Institute of Allergy & Infectious Diseases Mycoses Study Group [EORTC/MSG] Consensus Group definitions, endemic fungal infections per the EORTC/MSG Consensus Group definitions, other fungal infections, viral, bacterial & parasitic infections & vaccine dissemination) & special interest infections (actinomycosis, Legionella & mononucleosis-like toxoplasmosis).
Time Frame: From baseline to Week 52
Population: Participants in the SAS who had pEoI and were adjudicated by IRs
Measure: Number; unit: Number of events meeting criteria
Arm/Group | Tofacitinib 5 mg BID | Tofacitinib 10 mg BID
Number analyzed (Participants) | 4 | 4
Number of events meeting criteria | 1 | 1

27. Primary Outcome: Adjudicated Gastrointestinal (GI) Perforation Events
Description: Pre-specified GI perforation events were adjudicated by committees of external experts who were blinded to treatment assignment. The pEoI were identified via search of AE/SAE listings using the MedDRA GI Perforation SMQ. The IRs determined if the pEoI met the criteria for EoI classification based on whether a GI perforation occurred and if yes, the location within the GI tract, possible contributing medical conditions and/or concomitant medications.
Time Frame: From baseline to Week 52
Population: Participants in the SAS who had pEoI and were adjudicated by IRs
Measure: Number; unit: Number of events meeting criteria
Arm/Group | Tofacitinib 5 mg BID | Tofacitinib 10 mg BID
Number analyzed (Participants) | 0 | 2
Number of events meeting criteria |  | 2

28. Primary Outcome: Adjudicated Interstitial Lung Disease (ILD) Events
Description: Pre-specified ILD events were adjudicated by committees of external experts who were blinded to treatment assignment. pEoI were identified by searches of the clinical, safety & laboratory databases (AEs coded to the MedDRA ILD SMQ and events nominated by the study clinician or clinical lead). The IRs determined if the pEoI met the criteria for EoI classification by assessment of the ILD event (probably ILD, possible ILD, alternative diagnosis likely, other or insufficient information to classify).
Time Frame: From baseline to Week 52
Population: Participants in the SAS who had pEoI and were adjudicated by IRs
Arm/Group | Tofacitinib 5 mg BID | Tofacitinib 10 mg BID
Number analyzed (Participants) | 0 | 0

29. Secondary Outcome: Length of Hospitalizations Due to Crohn's Disease
Description: The length of hospitalizations due to Crohn's disease were recorded at every study visit.
Time Frame: From baseline to Week 52/follow-up
Population: SAS
Measure: Number; unit: Percentage of participnats
Arm/Group | Tofacitinib 5 mg BID | Tofacitinib 10 mg BID
Number analyzed (Participants) | 62 | 88
Percentage of participnats
  <3 days | 1.6 | 2.3
  3 to 6 days | 6.5 | 10.2
  7 to 10 days | 0 | 3.4
  > 10 days | 0 | 3.4

ADVERSE EVENTS:
Time Frame: SAEs were assessed from informed consent through and including 28 calendar days after last administration of study treatment. Non-SAEs were recorded from time of first dose of study treatment through last participant visit.
Description: The same event may appear as both an AE and an SAE. However, what is presented are distinct events. An event may be categorized as serious in 1 participant and as nonserious in another participant, or 1 participant may have experienced both a serious and nonserious event during the study.
Arm/Group | Tofacitinib 5 mg BID | Tofacitinib 10 mg BID
Serious Adverse Events (participants affected / at risk) | 5/62 | 14/88
Other Adverse Events (participants affected / at risk) | 42/62 | 58/88
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tofacitinib 5 mg BID (N=62) | Tofacitinib 10 mg BID (N=88)
Colon dysplasia (Gastrointestinal disorders) | 1 | 0
Crohn's disease (Gastrointestinal disorders) | 3 | 7
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 2
Chest pain (General disorders) | 1 | 0
Influenza like illness (General disorders) | 1 | 0
Pyrexia (General disorders) | 0 | 1
Biliary colic (Hepatobiliary disorders) | 0 | 1
Hypersensitivity (Immune system disorders) | 0 | 1
Anal abscess (Infections and infestations) | 0 | 1
Diarrhoea infectious (Infections and infestations) | 1 | 0
Pyelonephritis (Infections and infestations) | 1 | 0
Vulval abscess (Infections and infestations) | 0 | 1
Incisional hernia (Injury, poisoning and procedural complications) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 1 | 0
Perineal fistula (Reproductive system and breast disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0
C-reactive protein increased (Investigations) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Tofacitinib 5 mg BID (N=62) | Tofacitinib 10 mg BID (N=88)
Anaemia (Blood and lymphatic system disorders) | 3 | 4
Vertigo (Ear and labyrinth disorders) | 0 | 2
Abdominal distension (Gastrointestinal disorders) | 2 | 3
Abdominal pain (Gastrointestinal disorders) | 7 | 7
Abdominal pain upper (Gastrointestinal disorders) | 1 | 2
Anal fissure (Gastrointestinal disorders) | 1 | 2
Aphthous ulcer (Gastrointestinal disorders) | 1 | 3
Constipation (Gastrointestinal disorders) | 2 | 1
Crohn's disease (Gastrointestinal disorders) | 19 | 11
Diarrhoea (Gastrointestinal disorders) | 3 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 3
Flatulence (Gastrointestinal disorders) | 0 | 2
Food poisoning (Gastrointestinal disorders) | 2 | 0
Haematochezia (Gastrointestinal disorders) | 1 | 2
Haemorrhoids (Gastrointestinal disorders) | 0 | 4
Nausea (Gastrointestinal disorders) | 2 | 9
Proctalgia (Gastrointestinal disorders) | 1 | 2
Toothache (Gastrointestinal disorders) | 3 | 0
Vomiting (Gastrointestinal disorders) | 1 | 6
Chest pain (General disorders) | 2 | 2
Cyst (General disorders) | 2 | 0
Fatigue (General disorders) | 1 | 4
Pyrexia (General disorders) | 1 | 6
Bartholin's abscess (Infections and infestations) | 0/30 | 1/41
Bartholinitis (Infections and infestations) | 0/30 | 2/41
Cystitis (Infections and infestations) | 2 | 0
Folliculitis (Infections and infestations) | 0 | 2
Gastroenteritis (Infections and infestations) | 7 | 2
Herpes zoster (Infections and infestations) | 1 | 2
influenza (Infections and infestations) | 5 | 8
Nasopharyngitis (Infections and infestations) | 8 | 7
Oral herpes (Infections and infestations) | 3 | 0
Pharyngitis (Infections and infestations) | 2 | 0
Upper respiratory tract infection (Infections and infestations) | 2 | 2
Urinary tract infection (Infections and infestations) | 8 | 7
Vaginal infection (Infections and infestations) | 1/30 | 0/41
Vaginitis bacterial (Infections and infestations) | 0/30 | 1/41
Vulvovaginal candidiasis (Infections and infestations) | 0/30 | 1/41
Vulvovaginal mycotic infection (Infections and infestations) | 0/30 | 2/41
Blood alkaline phosphatase increased (Investigations) | 2 | 0
Blood creatine phosphokinase increased (Investigations) | 3 | 5
C-reactive protein increased (Investigations) | 2 | 0
Gamma-glutamyltransferase increased (Investigations) | 2 | 0
Lymphocyte count decreased (Investigations) | 1 | 2
Smear cervix abnormal (Investigations) | 1/30 | 0/41
Weight decreased (Investigations) | 2 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 2
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 2
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 0 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 | 8
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 4
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 | 2
Acrochordon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Headache (Nervous system disorders) | 1 | 2
Anxiety (Psychiatric disorders) | 0 | 3
Insomnia (Psychiatric disorders) | 2 | 0
Amenorrhoea (Reproductive system and breast disorders) | 0/30 | 1/41
Balanoposthitis (Reproductive system and breast disorders) | 1/32 | 0/47
Erectile dusfunction (Reproductive system and breast disorders) | 1/32 | 0/47
Oligomenorrhoea (Reproductive system and breast disorders) | 0/30 | 1/41
Testicular swelling (Reproductive system and breast disorders) | 0/32 | 1/47
Vulvovaginal pruritus (Reproductive system and breast disorders) | 0/30 | 1/41
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 2
Rash (Skin and subcutaneous tissue disorders) | 1 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less